CLINICAL TRIAL: NCT05131659
Title: Intervention-Induced Plasticity of Flexibility and Learning Mechanisms in ASD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: Georgetown University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Lauren Kenworthy, ASSOC CHIEF NEUROPSYCHOLOGY, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00015492; 1P50HD105328-01 (NIH)
Record Dates: First submitted 2021-09-30; First posted 2021-11-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Executive Dysfunction; Autism Spectrum Disorder; Adolescent Behavior
Keywords: Autism Spectrum Disorder; Executive Function; Intervention; MRI Scanning; Neuroimaging; Learning Mechanisms
MeSH Terms: conditions — Autism Spectrum Disorder; Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Executive function group therapy (Experimental)
  Interventions: Behavioral: Executive function group therapy

INTERVENTIONS:
Behavioral: Executive function group therapy — This executive function group therapy curriculum for adolescents uses cognitive behavioral therapy techniques, and focuses on key functions needed for adult success, such as: self-advocacy, flexibility, time management, motivation, goal setting, developing plans, monitoring progress. Guided practice begins with concrete interventionist support and moves to interventionist cueing, self-cueing, and finally automatic use of the skills without support.
  Other Names: Proprietary name: Unstuck & On Target (UOT:HS)

SUMMARY:
This project explores the association between learning and cognitive flexibility by testing whether a cognitive behavioral intervention designed to improve flexibility in ASD changes learning and associated neural activation using model-based functional magnetic resonance imaging (m-fMRI). The study proposes that variability in learning mechanisms is associated with behavioral flexibility and explains differences in adaptive and treatment outcomes. The study employs a longitudinal case-controlled design in 60 14-18 year old youth with ASD at 3 time-points 8 months apart, each including m-fMRI during learning and behavioral measurement of executive and adaptive function. Aim 1 tests the hypothesis that individual variation in learning biases and their neural correlates predicts behavioral flexibility and is stable over time. Aim 2 tests plasticity of learning mechanisms induced by a cognitive-behavioral intervention for flexibility. Aim 3 tests hypothesis about intervention-induced plasticity of neural functional connectivity.

ELIGIBILITY:
Inclusion Criteria:

1. 14-18 years of age inclusive
2. Full scale IQ > 80 on a standardized IQ test, either confirmed through educational testing within the last two years or confirmed by the Wechsler Abbreviated Scale of Intelligence (WASI-2) administered by research personnel. If current IQ testing (FSIQ) is not interpretable based on discrepancies between verbal and perceptual skills, we will use the best available verbal IQ estimate.
3. Broad ASD diagnosis according to Diagnostic Statistical Manual, fifth edition (DSM-5) criteria established by parent report of prior clinical diagnosis and confirmed by meeting cutoff criteria on the Social Communication Questionnaire (i.e., raw score > 11) or the Autism Diagnostic Observation Schedule-2 (ADOS-2), Module 4 (total score ≥7).
4. Intact or corrected hearing and vision.
5. Parents/guardians speak and read English with sufficient fluency for completion of consent forms and informant questionnaires; youth participants will use/understand English as a primary or secondary language with sufficient fluency to engage effectively in executive function group therapy conducted in English, and for valid administration of neuropsychological and behavioral measures.

Exclusion Criteria:

1. Presence of a known medical condition in the participant that would interfere with his/her ability to participate in the study.
2. To preserve the integrity of the neuroimaging data, participants will be excluded if they have a history of neurological disorder, such as an established epilepsy diagnosis, significant brain trauma, hydrocephalus, central nervous system infection, or stroke.
3. Contraindications for MRI such as metal implants, dental braces, pregnancy (determined by parent or self-report).

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Executive Function Challenge Task (EFCT) Scores | 8-12 months before intervention, at start of intervention, 8-12 months after intervention begins
  The EFCT is an objective and ecologically valid task developed by our research team to assess flexibility and planning skills in a social context conducted by a trained research staff member masked to treatment condition. The EFCT uses a standardized, semi-structured protocol which does not provide explicit rules for completing the tasks to mimic the implicit, unspoken, unstructured expectations in everyday life. The EFCT consists of challenges across several activities and responses are scored on a 3-point scale for each task. The scale (0-good, 1-intermediate, 2-poor performance) has task-specific behavioral markers to guide scoring.
Change in Neural Response During Prototype Learning Task Outcomes | 8-12 months before intervention, at start of intervention, 8-12 months after intervention begins
  The Prototype Task measures learning of abstract representations in the visual domain. The task requires classification into two categories of visual exemplars characterized by a number of features (e.g., cartoon fish with features such as a particular eye shape, fins, body shape etc.) for training with feedback. Following training, generalization of learned information is tested on exemplars that are similar to training items but have never been presented before. Participants perform the generalization phase in an MRI scanner for measurement of brain activation. Learning of abstract visual representation (e.g., prototype learning) on this task is indicated by engagement of medial prefrontal cortex (mPFC)

SECONDARY OUTCOMES:
Change in Adaptive Behavior Assessment System, Third Edition (ABAS-3) scores | 8-12 months before intervention, at start of intervention, 8-12 months after intervention begins
  Adaptive behavior will be measured via parent-report on the Adaptive Behavior Assessment System, Third Edition (ABAS-3). The ABAS-3 is a well-validated parent report measure that assesses practical, everyday skills needed to effectively and independently take care of oneself and interact with others across the lifespan.

OTHER OUTCOMES:
Change in Prototype Task Performance: Learning Strategy Scores | 8-12 months before intervention, at start of intervention, 8-12 months after intervention begins
  Generalization phase learning can be characterized by strategy using computational modeling. Two models are tested; 1. learning from having abstracted information that is prototypical of the category (e.g., family of fish as described above); 2. Learning from matching exemplar information to training phase
Change in Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2) Scores | 8-12 months before intervention, at start of intervention, 8-12 months after intervention begins, 8-12 months after intervention ends
  The BRIEF-2 is a well-established self-report measure of real-world EF skills, with the Shift subscale measuring cognitive flexibility.
Change in Dimensional Change Card Sort Test (DCCS) Scores | 8-12 months before intervention, at start of intervention, 8-12 months after intervention begins
  The Dimensional Change Card Sort Test (NIH Toolbox) is a 4-minute, standard lab-based task for assessing cognitive flexibility in terms of set-shifting. Participants are required to sort a series of bivalent cards first according to one dimension (e.g., color) and then according to another (e.g., shape). It is normed from ages 4-85
Change in Flexibility Scale Scores | 8-12 months before intervention, at start of intervention, 8-12 months after intervention begins, 8-12 months after intervention ends
  The Flexibility Scale (FS) is a 27-item measure assessing five categories related to flexibility: routines and rituals, transitions/change, special interests, social flexibility and generativity
Change in CVLT-C Scores | 8-12 months before intervention, at start of intervention, 8-12 months after intervention begins
  California Verbal Learning Test Children's Version (CVLT-C) is used to assess verbal learning and memory through an everyday memory task in which the child is asked to recall a list. The measure is for children and adolescents 5 through 16.11 years
Change in CVLT-3 Scores | 8-12 months before intervention, at start of intervention, 8-12 months after intervention begins
  California Verbal Learning Test Adolescent and Adult Version (CVLT-3) is used to assess verbal learning and memory through an everyday memory task in which the individual is asked to recall a list. The measure is for Individuals between 16-90 years old
Change in ASC - ASD Scores | 8-12 months before intervention, at start of intervention, 8-12 months after intervention begins, 8-12 months after intervention ends
  The Anxiety Scale for Children- ASD (ASC-ASD) is a 24 item self-report anxiety questionnaire, with four sub-scales: Separation Anxiety (SA), Uncertainty (U), Performance Anxiety (PA) and Anxious Arousal (AA), for use with young people aged between 8-16 years with a diagnosis of autism spectrum disorder (ASD).
Change in AIR-SDS Scores | 8-12 months before intervention, at start of intervention, 8-12 months after intervention begins, 8-12 months after intervention ends
  The AIR Self-Determination scale (AIR-SDS) produces a profile of the student's level of self-determination, identifies areas of strength and areas needing improvement, identifies specific educational goals that can be incorporated into the student's individualized education plan (IEP). The measure examines two broad self-determination components. Capacity refers to the student's knowledge, abilities, and perceptions that enable them to be self-determined. Opportunity refers to the student's chances to use their knowledge and abilities
Change in PRAS-ASD Scores | 8-12 months before intervention, at start of intervention, 8-12 months after intervention begins, 8-12 months after intervention ends
  Parent-Rated Anxiety Scale for Autism Spectrum Disorder (PRAS-ASD) is 25-item measure for anxiety. This is a reliable and valid measure that can be used to assess severity of anxiety in youth with ASD and evaluate change with treatment
Change in Rey Complex Figure Test and Recognition Trial Scores | 8-12 months before intervention, at start of intervention, 8-12 months after intervention begins
  Rey Complex Figure Test and Recognition Trial (RCFT) tests visuospatial constructional ability and visuospatial memory using the "complex figure." The RCFT consists of four separate tasks and is scored using specific criteria developed for scoring the accuracy and placement of individual units of the complex figure
Change in BDI-II Scores | 8-12 months before intervention, at start of intervention, 8-12 months after intervention begins, 8-12 months after intervention ends
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's National Hospital, Washington D.C., District of Columbia
  - Georgetown University, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT05131659/Prot_SAP_000.pdf